CLINICAL TRIAL: NCT00471523
Title: Clomiphene Citrate Versus Metformin as First-Line Approach for the Treatment of Anovulation in Infertile Patients With Polycystic Ovary Syndrome
Brief Title: Treatment of Anovulatory Infertility in PCOS Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-2006
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-05

CONDITIONS: Infertility; Polycystic Ovary Syndrome; Anovulation
Keywords: Anovulation; Clomiphene citrate; Infertility; Metformin; PCOS; Treatment
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome; Anovulation | interventions — Clomiphene; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clomiphene citrate
Drug: Metformin

SUMMARY:
Clomiphene citrate (CC) and metformin are two effective drugs used to induce ovulation in patients with polycystic ovary syndrome (PCOS), even if it is still unclear which compound between them should be initially administered. The aim of the study will be to compare in a clinical setting the efficacy of CC and metformin as first-line approaches for treating anovulation in infertile PCOS patients.

DETAILED DESCRIPTION:
Eighty infertile anovulatory patients with PCOS will be allocated in two body mass index (BMI)- and age-matched groups (experimental and control groups).

Forty patients will receive the experimental treatment consisting of six months of 1700 mg/day metformin administration (experimental group), whereas other forty patients will receive CC administered using a traditional incremental-doses protocol (control group). In both groups, patients who will ovulate under treatment will continue the therapy for a total of six months.

During the study, the clinical and reproductive outcomes, and the adverse experience will be evaluated in each patient.

ELIGIBILITY:
Inclusion Criteria:

* Anovulatory infertility related to polycystic ovary syndrome

Exclusion Criteria:

* Neoplastic, metabolic, hepatic, and cardiovascular disorders or other concurrent medical illnesses
* Hypothyroidism, hyperprolactinemia, Cushing's syndrome, and non-classical congenital adrenal hyperplasia
* Current or previous (within the last six months) use of oral contraceptives, glucocorticoids, antiandrogens, ovulation induction agents, antidiabetic and anti-obesity drugs or other hormonal drugs.
* Organic pelvic diseases
* Previous pelvic surgery
* Suspected peritoneal factor infertility
* Tubal or male factor infertility or sub-fertility

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2006-05; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 10 months

SECONDARY OUTCOMES:
Ovulation rate | 6 months
Abortion rate | 10 months
Time to first pregnancy | 10 months
Adverse events | 10 months
N. pregnancies/n. ovulatory cycles | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics & Gynecology, University "Magna Graecia" of Catanzaro; Achille Tolino, MD, Principal Investigator — Department of Obstetrics & Gynecology, University "Federico II" of Naples; Francesco Orio, MD, Principal Investigator — Department of Endocrinology, University "Federico II" of Naples
Locations (1):
- "Pugliese Hospital", Catanzaro, CZ, Italy

REFERENCES:
- [Background] Palomba S, Orio F Jr, Falbo A, Manguso F, Russo T, Cascella T, Tolino A, Carmina E, Colao A, Zullo F. Prospective parallel randomized, double-blind, double-dummy controlled clinical trial comparing clomiphene citrate and metformin as the first-line treatment for ovulation induction in nonobese anovulatory women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2005 Jul;90(7):4068-74. doi: 10.1210/jc.2005-0110. Epub 2005 Apr 19. PMID 15840746
- [Background] Palomba S, Orio F Jr, Falbo A, Russo T, Tolino A, Zullo F. Effects of metformin and clomiphene citrate on ovarian vascularity in patients with polycystic ovary syndrome. Fertil Steril. 2006 Dec;86(6):1694-701. doi: 10.1016/j.fertnstert.2006.05.035. Epub 2006 Oct 30. PMID 17074337
- [Background] Palomba S, Orio F, Zullo F. Ovulation induction in women with polycystic ovary syndrome. Fertil Steril. 2006 Jul;86 Suppl 1:S26-7. doi: 10.1016/j.fertnstert.2006.03.018. PMID 16798282
- [Background] Palomba S, Russo T, Orio F Jr, Falbo A, Manguso F, Sammartino A, Tolino A, Colao A, Carmina E, Zullo F. Uterine effects of clomiphene citrate in women with polycystic ovary syndrome: a prospective controlled study. Hum Reprod. 2006 Nov;21(11):2823-9. doi: 10.1093/humrep/del267. Epub 2006 Jul 10. PMID 16835214
- [Derived] Palomba S, Falbo A, Orio F Jr, Tolino A, Zullo F. Efficacy predictors for metformin and clomiphene citrate treatment in anovulatory infertile patients with polycystic ovary syndrome. Fertil Steril. 2009 Jun;91(6):2557-67. doi: 10.1016/j.fertnstert.2008.03.011. Epub 2008 Apr 28. PMID 18440534